CLINICAL TRIAL: NCT01160107
Title: A Multicenter, Open Label Study Of Oral Revlimid And Prednisone (Rp) Followed By Oral Revlimid Melphalan And Prednisone (Mpr) In Newly Diagnosed Elderly Multiple Myeloma Patients
Brief Title: Revlimid And Prednisone Followed By Revlimid, Melphalan And Prednisone In Multiple Myeloma Patients
Acronym: RP_MPR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione EMN Italy Onlus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RV-MM-PI-302; 2007-007616-28 (EudraCT Number)
Record Dates: First submitted 2010-07-09; First posted 2010-07-12 (Estimated); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Multiple Myeloma
Keywords: Diagnosis; Elderly Patients; Imids; Chemotherapy
MeSH Terms: conditions — Multiple Myeloma; Disease | interventions — Lenalidomide; Prednisone; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RP followed MPR (Experimental)
  Interventions: Drug: RP followed by MPR

INTERVENTIONS:
Drug: RP followed by MPR — Induction (4 cycles):Lenalidomide 25 mg/die for 21 days followed by a 7 days rest period and Prednisone at 50 mg three times a week continuously . Consolidation (6 cycles): Melphalan 2 mg three times a week, Prednisone 50 mg three times a week, and Lenalidomide 15 mg/die for 21 days followed by a 7 days rest period. According to the results of the first stage the decisions are as follows: 1. Starting a second stage, at the same dose of lenalidomide for MPR cycles, if grade 3-4 adverse events are 25-50% and PR > 50%; 2. The study stop (if PR <40% and grade 3-4 adverse events >25-30%) 3. A new first stage may be started: - Lenalidomide 20 mg/die if grade 3-4 adverse events are < 25-30%, independently from efficacy; - Lenalidomide 10 mg/die if grade 3-4 adverse events are > 50% and PR rate > 50%. Maintenance: Lenalidomide 10 mg/day from day 1 to 21, followed by a 7-day rest period and Prednisone 25 mg three times a week.Each cycle will be repeated every 28 days, until PD.
  Other Names: Revlimid; Prednisone; Melphalan

SUMMARY:
This study will determine whether the association of Revlimid and Prednisone (RP) as induction treatment followed by Revlimid, Melphalan and Prednisone (MPR) as consolidation treatment is safe and induce a significant rate of PR (and CR) in newly diagnosed elderly MM patients.

DETAILED DESCRIPTION:
This phase II study is a multicenter, open label trial designed to determine whether the association of Revlimid and Prednisone (RP) as induction treatment followed by Revlimid, Melphalan and Prednisone (MPR) as consolidation treatment is safe and induce a significant rate of PR (and CR) in newly diagnosed elderly MM patients.

This study consists of 3 phases for each study subject: Pre-treatment, Treatment, long-term follow-up (LTFU).

Pre-treatment period: after providing written informed consent, patients will undergo screening for protocol eligibility as outlined in the Schedule of Study Assessments.

Treatment period: includes induction, consolidation and maintenance.

Induction regimen:Patients will start induction treatment with association of Lenalidomide and Prednisone (RP).

Consolidation regimen After the completion of the 4 RP cycles therapy will continue with the MPR association:·

According to the results after the first stage the decisions are as follows: 1. The study may continue to a second stage, at the same dose of lenalidomide of MPR cycles, if grade 3-4 adverse events are 25-50% and PR > 50%;

2. The study may be stopped (if PR < 40% and grade 3-4 adverse events > 25-30%)

3. A new first stage may be started:

* At an increase dose of Lenalidomide administered in advanced MPR cycles if grade 3-4 adverse events are < 25-30%, independently from efficacy;
* At a reduced dose of Lenalidomide administered in advanced MPR cycles if grade 3-4 adverse events are > 50% and PR rate > 50%

Maintenance: Within 3 months from the last MPR cycle, therapy will continue with RP as maintenance.

Each cycle will be repeated every 28 days, until PD.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 65 years of age or older at the time of signing the informed consent.
* Patient is, in the investigator(s) opinion willing and able to comply with the protocol requirements.
* Patient has given voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to their future medical care.
* Male patient agrees to use an acceptable method for contraception (i.e., condom or abstinence) during study drug therapy (including dose interruption) and for 4 weeks after discontinuation of lenalidomide therapy.
* Female patient is either post-menopausal for 24 consecutive months or surgically sterilised or agree to continuous abstinence from heterosexual sexual contact or willing to use two acceptable method of birth control at the same time (one highly effective method and one additional effective method)(Highly Effective Methods: Intrauterine device -IUD-; Hormonal -birth control pills, injections, implants-; tubal ligation; partner's vasectomy; Additional Effective Methods: Latex condom; Diaphragm; Cervical Cap) for 4 weeks prior to beginning study drug therapy, during study drug therapy (including dose interruption) and for 4 weeks after discontinuation of lenalidomide therapy.
* Patient was a newly diagnosed multiple myeloma based on standard criteria
* Patient has measurable disease, defined as follows: - Secretory myeloma: any quantifiable serum monoclonal protein value (generally, but not necessarily, greater than 1 g/dL of IgG M-Protein and greater than 0.5 g/dL of IgA M-Protein) and, where applicable, urine light-chain excretion of >200 mg/24 hours; - Non-secretory myeloma: > 30% plasma cells in the bone marrow and at least one plasmacytoma > 2 cm as determined by clinical examination or applicable radiographs (i.e., MRI or CT scan).
* Patient has a Karnofsky performance status ≥ 50%.
* Patient has a life-expectancy >3 months.

Exclusion Criteria:

* Any serious medical condition, laboratory abnormality or psychiatric illness that prevented the subject from signing the informed consent form or placed the subjects at unacceptable risk.
* Previous treatment with anti-myeloma therapy (does not include radiotherapy, bisphosphonates, or a single short course of steroid; < to the equivalent of dexamethasone 40 mg/day for 4 days).
* Pregnant or lactating females
* Known positive for HIV or active infectious hepatitis type A, B or C

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 46 (Actual)
Dates: Start 2008-07 (Actual); Primary Completion 2012-08 (Actual); Study Completion 2022-12-22 (Actual)

PRIMARY OUTCOMES:
RP as induction followed by MPR as consolidation treatment is safe and induce a significant rate of PR (and CR) | Approximately 24 months
  Determine whether the association of RP as induction followed by MPR as consolidation treatment is safe and induce a significant rate of PR (and CR) in elderly patients with newly diagnosed multiple myeloma.

SECONDARY OUTCOMES:
Determine the progression free survival (PFS), overall survival (OS) and whether responses obtained with RP - MPR treatment, are associated with a prolongation of PFS, in comparison with non-responding patients. | Approximately 24 months
  The secondary objectives of this study are:
  * To determine progression free survival (PFS)
  * To determine overall survival (OS)
  * To determine whether responses obtained with RP - MPR treatment, are associated with a prolongation of PFS, in comparison with non-responding patients.

CONTACTS AND LOCATIONS:
Overall Officials: Mario Boccadoro, MD, Principal Investigator — S.C. Ematologia U - AOU CITTA' DELLA SALUTE E DELLA SCIENZA DI TORINO